CLINICAL TRIAL: NCT01715090
Title: Web-based Insulin Titration: Improving Diabetes Care in the Netherlands. An Efficacy Study.
Brief Title: Web-based Insulin Titration - An Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 40248.018.12
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based insulin titration (Experimental): An online web-based insulin titration algorithm to guide patients in self-titration
  Interventions: Device: Web-based insulin titration
- Standard care (No Intervention)

INTERVENTIONS:
Device: Web-based insulin titration
  Other Names: PANDIT
  Arms: Web-based insulin titration

SUMMARY:
The main objective of the study is to determine whether an intensive web-based titration system, called PANDIT (Patient Assisting Net-based Diabetes Insulin Titration), is effective in improving glycaemic control in patients with diabetes mellitus type 2 using a basal insulin, compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 80 years
* Type 2 diabetes mellitus (diagnosed clinically) for ≥ 6 months
* Once daily basal insulin therapy usage
* No restriction on HbA1c or FPG
* BMI < 40 kg/m2
* Ability to read and understand the Dutch language
* Familiarity with the Internet and use of a mobile phone
* Ability and willingness to adhere to the protocol
* Ability and willingness to use a web-based insulin self-titration system
* Confirmed written consent

Exclusion Criteria:

* Type 1 diabetes
* Use of systemic corticosteroid in the last three months
* Recurrent severe hypoglycaemia or hypoglycaemic unawareness
* Active proliferative diabetic retinopathy
* Any clinically significant disease or disorder
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Working in night shifts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c | Change from baseline after 13 weeks and after 26 weeks

SECONDARY OUTCOMES:
Quality of life and treatment satisfaction | Change from baseline after 13 weeks and after 26 weeks
Total contact time with study staff (and the PANDIT system, if applicable) | After 26 weeks
Proportion of subjects who reach the target of HbA1c < 7.0% | After 26 weeks
Mean change in fasting plasma glucose | Change from baseline after 13 weeks and after 26 weeks
Overall incidence and rate of hypoglycaemia (mild hypoglycaemia, probable hypoglycaemia, severe hypoglycaemia and relative hypoglycaemia) | After 26 weeks
Frequency of the usage of PANDIT among patients | After 26 weeks
Detection of important factors for patient compliance to internet-based self-care interventions | After 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frits Holleman, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Result] Simon AC, Holleman F, Hoekstra JB, De Clercq PA, Lemkes BA, Hermanides J, Peek N. Development of a web-based decision support system for insulin self-titration. Stud Health Technol Inform. 2011;169:103-7. PMID 21893723
- [Result] Simon AC, Holleman F, Gude WT, Hoekstra JB, Peek N. Safety of a web-based insulin titration system for patients with type 2 diabetes mellitus - pilot study. Stud Health Technol Inform. 2012;180:731-5. PMID 22874288
- [Result] Gude WT, Simon AC, Peute LW, Holleman F, Hoekstra JB, Peek N, Jaspers MW. Formative usability evaluation of a web-based insulin self-titration system: preliminary results. Stud Health Technol Inform. 2012;180:1209-11. PMID 22874403